CLINICAL TRIAL: NCT03639623
Title: A Phase 2A, Single Center, Open-label, Single-arm, 24-week Study to Evaluate the Safety, Tolerability and Efficacy of Saroglitazar Magnesium 4 mg in Liver Transplant Recipients With Nonalcoholic Fatty Liver Disease (EVIDENCES VIII)
Brief Title: Safety, Tolerability, and Efficacy of Saroglitazar Mg 4 mg in Liver Transplant Recipients With Nonalcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARO.17.010
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Liver Transplant; Complications; NAFLD
Keywords: Peroxisome proliferator-activated receptors; NAFLD; NASH; Post Transplant Metabolic Syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — saroglitazar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Saroglitazar Magnesium 4 mg (Experimental): Saroglitazar Magnesium tablet once daily in the morning 60 minutes before breakfast
  Interventions: Drug: Saroglitazar

INTERVENTIONS:
Drug: Saroglitazar — Saroglitazar magnesium 4 mg tablet once daily (OD) in the morning 60 minutes before breakfast without food
  Other Names: Not any

SUMMARY:
This is a phase 2A, single center, open-label, single-arm, 24-week study to evaluate the safety, tolerability and efficacy of Saroglitazar Magnesium 4 mg in liver transplant recipients with NAFLD.

DETAILED DESCRIPTION:
This is a phase 2A, single center, open-label, single-arm, 24-week study to evaluate the safety, tolerability and efficacy of Saroglitazar Magnesium 4 mg in liver transplant recipients with NAFLD.

The study will be conducted over a period of up to 33 weeks and will include 5 weeks screening, a 24 week treatment period and 4 week follow-up period. The primary end point of the study is to assess the safety of Saroglitazar Magnesium 4 mg in liver transplant recipients with NAFLD over 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Males or females, 18 to 75 years of age.
* Patients who are at least 6 months post-transplant for nonalcoholic steatohepatitis (NASH) or cryptogenic cirrhosis thought to be secondary to NASH are eligible for enrolment.
* The presence of NAFLD determined by Magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF) prior to enrollment.
* Patients with ≤20% variance in the levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin between Visit 1 and Visit 1.1.
* History of medical compliance with immunosuppression.
* Female subjects of non-child bearing potential or on highly effective contraception. For male subjects with female partners of childbearing potential, willing to follow highly effective contraception measures during the study, either by the male participant or his female partner or both.

Exclusion Criteria:

* Pregnant or lactating females.
* Patient with abnormal transaminases due to secondary intercurrent illness.
* Patients with bile duct strictures.
* Other causes of chronic liver disease after liver transplantation including autoimmune, viral, and alcoholic liver disease.
* Graft cirrhosis as defined by:

  1. Cirrhosis on historical liver biopsy.
  2. Evidence of cirrhosis on imaging including portal venous collaterals.
  3. Prior history of decompensated liver disease including ascites, hepatic encephalopathy or variceal bleeding.
  4. Evidence of esophageal varices on prior endoscopy.
* Body mass index (BMI) <18 kg/m².
* Subjects with change in body weight >5% in the 3 months prior to enrollment.
* Subjects requiring corticosteroid or anticoagulation therapy.
* History of myopathies or evidence of active muscle diseases.
* Unstable cardiovascular disease.
* History of bladder disease and/or hematuria or has current hematuria unless due to a urinary tract infection.
* Active malignancy post-liver transplantation.
* History of malignancy in the past 5 years and/or active neoplasm.
* History of chronic rejection of liver transplant graft.
* Acute cellular rejection of liver transplant graft within the past 6 months.
* Evidence of Acute cellular rejection (ACR) or chronic rejection (CR) or alternative etiologies to NAFLD.
* Poorly controlled diabetes as defined by an HbA1c >8.5% within the past 6 months.
* History of excessive alcohol intake.
* Subject tests positive for a urine drug screen.
* Subject has a history of chronic (uncontrolled) pain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deven Parmar, MD FCP, Study Director — Zydus Therapeutics Inc.
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhati C, Idowu MO, Sanyal AJ, Rivera M, Driscoll C, Stravitz RT, Kohli DR, Matherly S, Puri P, Gilles H, Cotterell A, Levy M, Sterling RK, Luketic VA, Lee H, Sharma A, Siddiqui MS. Long-term Outcomes in Patients Undergoing Liver Transplantation for Nonalcoholic Steatohepatitis-Related Cirrhosis. Transplantation. 2017 Aug;101(8):1867-1874. doi: 10.1097/TP.0000000000001709. PMID 28296807
- [Result] Siddiqui MS, Parmar D, Shaikh F, Forsgren M, Patel S, Bui AT, Boyett S, Patel V, Sanyal AJ. Saroglitazar improves nonalcoholic fatty liver disease and metabolic health in liver transplant recipients. Liver Transpl. 2023 Sep 1;29(9):979-986. doi: 10.1097/LVT.0000000000000110. Epub 2023 Feb 28. PMID 36847136
- See also: Bhati C, Idowu MO, Sanyal AJ. Long-term Outcomes in Patients Undergoing Liver Transplantation for Nonalc — http://pubmed.ncbi.nlm.nih.gov/28296807/
- See also: Siddiqui MS, Parmar D, Shaikh F, Forsgren M, Patel S, Bui AT, Boyett S, Patel V, Sanyal AJ. Saroglitazar improves nonalcoholic fatty liver disease and metabolic health in liver transplant recipients — http://pubmed.ncbi.nlm.nih.gov/36847136/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saroglitazar Magnesium 4 mg
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 36.8 (6.77)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Assessed by CTCAE
Description: Safety measured by adverse events, vital signs, physical exams, body weight, electrocardiograms (ECGs) and lab results (including hematology, chemistry and urinalysis)
Time Frame: 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 20
Participants | 12

2. Secondary Outcome: Hepatic Fat
Description: Changes in hepatic fat as determined by MRI-PDFF from baseline to end-of-treatment (EOT)
Time Frame: Baseline and week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percentage of hepatic fat
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
percentage of hepatic fat | -3.17 (5.82)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.053, paired t-test

3. Secondary Outcome: Liver Stiffness
Description: Changes in Liver stiffness as determined by MRE from baseline to end-of-treatment (EOT) Liver stiffness is a measure of a mechanical property of tissue (stiffness). This can be measured non-invasively by MR elastography, a technique that involves applying an external vibration to the abdomen and measuring the progression of shear waves through the underlying liver using MRI.
Time Frame: Baseline and Week 24
Population: Modified-in-to-treat population
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
kPa | 0.01 (0.34)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.958, paired t-test

4. Secondary Outcome: Frequently Sampled Intravenous Glucose Tolerance Test (Insulin Resistance Marker)
Description: Changes in frequently sampled intravenous glucose tolerance test (FSIVGTT) from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
mg/dL | -22.68 (29.99)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.011, paired t-test

5. Secondary Outcome: Glycosylated Hemoglobin (Insulin Resistance Marker)
Description: Changes in glycosylated hemoglobin (HbA1c) from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
percentage of glycosylated hemoglobin | -0.11 (0.57)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.454, paired t-test

6. Secondary Outcome: Fructosamine (Insulin Resistance Marker)
Description: Changes in fructosamine from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
µmol/L | -10.90 (28.13)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.154, paired t-test

7. Secondary Outcome: Serum Liver Enzymes
Description: Changes in serum liver enzymes from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified-intent-to-treat population
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
U/L
  Change in ALT | -9.10 (23.23)
  Change in AST | 3.90 (17.56)
  Change in ALP | -42.80 (22.07)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: ALT; Test type: Other; p = 0.125, paired t-test
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: AST; Test type: Other; p = 0.375, paired t-test
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: ALP; Test type: Other; p < 0.001, paired t-test

8. Secondary Outcome: Serum Liver Enzymes; Bilirubin
Description: Changes in bilirubin from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified-intent-to-treat population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
mg/dL | -0.08 (0.16)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.054, paired t-test

9. Secondary Outcome: Serum Lipids
Description: Changes in serum lipids from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified Intent-to-treat population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
mg/dL
  Change in Total Cholesterol | -5.50 (20.74)
  Change in Triglycerides | -43.20 (47.92)
  Change in Non-HDL-C | -6.20 (17.31)
  Change in HDL-C | 0.20 (10.27)
  Change in HDL-C Subclass 2 | -5.30 (9.39)
  Change in HDL-C Subclass 3 | 5.10 (5.75)
  Change in LDL-C | 2.90 (19.40)
  Change in VLDL-C | -8.50 (9.49)
  Change in VLDL concentration | -6.60 (13.63)
  Change in Small dense LDL-C | -4.29 (5.17)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Outcome variable: Total Cholesterol; Test type: Other; p = 0.378, paired t-test
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: Triglyceride; Test type: Other; p = 0.010, paired t-test
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: Non-HDL-C; Test type: Other; p = 0.264, paired t-test
Statistical Analysis 4: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: HDL-C; Test type: Other; p = 0.954, paired t-test
Statistical Analysis 5: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: HDL-C Subclass 2; Test type: Other; p = 0.127, paired t-test
Statistical Analysis 6: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: HDL-C Subclass 3; Test type: Other; p = 0.029, paired t-test
Statistical Analysis 7: Comparison: Saroglitazar Magnesium 4 mg; Outcome variable: LDL-C; Test type: Other; p = 0.630, paired t-test
Statistical Analysis 8: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: VLDL-C; Test type: Other; p = 0.010, paired t-test
Statistical Analysis 9: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: VLDL concentration; Test type: Other; p = 0.160, paired t-test
Statistical Analysis 10: Comparison: Saroglitazar Magnesium 4 mg; Small dense LDL-C; Test type: Other; p = 0.020, paired t-test

10. Secondary Outcome: Small Dense Low-density Lipoprotein (Atherogenic Lipoprotein)
Description: Changes in small dense low-density lipoprotein (sdLDL) from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
nmol/L | 51.40 (248.45)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.529, paired t-test

11. Secondary Outcome: LDL Size (Atherogenic Lipoprotein)
Description: Changes in LDL size from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
nm | 0.17 (0.61)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: LDL Size; Test type: Other; p = 0.403, paired t-test

12. Secondary Outcome: LDL Concentration (Atherogenic Lipoprotein)
Description: Changes in LDL concentration from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
nmol/L | 21.70 (155.44)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.669, paired t-test

13. Secondary Outcome: Very Low-density Lipoprotein (Atherogenic Lipoprotein)
Description: Changes in subtypes of very low-density lipoprotein (VLDL) from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
nmol/L
  Change in VLDL chylomicron particles | -20.22 (22.92)
  Change in Large VLDL chylomicron particles | -2.20 (2.19)
  Change in Medium VLDL particles | -13.24 (19.47)
  Change in Small VLDL particles | -4.79 (14.53)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: VLDL chylomicron particles; Test type: Other; p = 0.021, paired t-test
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: Large VLDL chylomicron particles; Test type: Other; p = 0.011, paired t-test
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: Medium VLDL particles; Test type: Other; p = 0.060, paired t-test
Statistical Analysis 4: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: Small VLDL particles; Test type: Other; p = 0.324, paired t-test

14. Secondary Outcome: Very Low-density Lipoprotein Chylomicron Triglyceride (Atherogenic Lipoprotein)
Description: Changes in VLDL chylomicron triglyceride from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
mg/dL | -40.70 (39.77)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.010, paired t-test

15. Secondary Outcome: High-density Lipoprotein (Atherogenic Lipoprotein)
Description: Changes in high-density lipoprotein (HDL) from baseline to EOT
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
µmol/L | 1.82 (4.67)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Test type: Other; p = 0.249, paired t-test

16. Secondary Outcome: Change in Metabolic Flexibility; Time to Peak RQ
Description: Metabolic flexibility was measured via a whole room calorimeter (i.e. respiration chamber). The CO2 production and O2 consumption were recorded every minute for a total of 18 hours while study participants were in the respiration chamber on baseline and Week 24. Metabolic flexibility was quantified by measuring whole-body CO2 production relative to O2 consumption or respiratory quotient (RQ). The RQ oscillates between 0.7 and 1.0, which is indicative of either predominantly fatty acid or carbohydrate oxidation, respectively.
  The time to maximal carbohydrate consumption is measured by the time it takes to reach peak RQ after a standardized meal, whereas maximal carbohydrate consumption is measured at the peak of RQ vs. time curve. Next, the transition from maximal carbohydrate consumption to maximal fatty acid consumption is measured from peak RQ to lowest RQ. Finally, fasting biofuel utilization is measured in the fasting state and represents predominantly fatty acid oxidation.
Time Frame: Baseline and Week 24
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 15
minutes | -53.2 (78.0)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Time to peak RQ; Test type: Other; p = 0.0193, paired t-test

17. Secondary Outcome: Quality of Life (SF-36 Health Survey)
Description: Change in Quality of life score from baseline to EOT The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the PCS and mental composite t-score (MCS). The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as the worst health status
Time Frame: Baseline and Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 17
score on a scale
  Physical Component Score | -0.10 (7.54)
  Mental Component Score | 2.63 (8.45)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: Physical component score; Test type: Other; p = 0.960, paired t-test
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg; Outcome Variable: Mental component score; Test type: Other; p = 0.249, paired t-test

18. Secondary Outcome: Peak Plasma Concentration [Cmax]
Description: Pharmacokinetics of Saroglitazar following first and last dose.
Time Frame: PK Sampling time points: Day 1 and Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
ng/mL
  first dose (Day 1) | 174.783 (53.673)
  last dose (Week 24) | 115.687 (62.680)

19. Secondary Outcome: Time to Reach Peak Plasma Concentration [Tmax]
Description: Pharmacokinetics of Saroglitazar following first and last dose
Time Frame: PK Sampling time points: Day 1 and Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
hours
  First dose (Day 1) | 1.010 [1.000 to 3.000]
  Last dose (Week 24) | 2.500 [0.500 to 4.000]

20. Secondary Outcome: Area Under Plasma Concentration vs. Time Curve Till the Last Time Point [AUC0-t]
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Day 1 visit at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: (ng/mL)*(hr)
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
(ng/mL)*(hr) | 689.550 (380.816)

21. Secondary Outcome: Area Under Plasma Concentration vs. Time Curve Extrapolated to the Infinity [AUC0-∞]
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Day 1 visit at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: (ng/mL)*(hr)
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
(ng/mL)*(hr) | 698.354 (386.372)

22. Secondary Outcome: Area Under Plasma Concentration vs. Time Curve in a 24 h Dosing Interval [AUCtau]
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Day 1 and Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: (ng/mL)*(hr)
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
(ng/mL)*(hr)
  First dose (Day 1) | 689.504 (380.751)
  Last dose (Week 24) | 805.178 (513.106)

23. Secondary Outcome: Elimination Rate Constant [λz]
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Day 1 and Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
L/hour
  First dose (Day 1) | 0.167 (0.020)
  last dose (Week 24) | 0.159 (0.024)

24. Secondary Outcome: Elimination Half-life [t1/2]
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Day 1 and Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
hour
  First dose (Day 1) | 4.199 (0.479)
  Last dose (Week 24) | 4.442 (0.612)

25. Secondary Outcome: Apparent Volume of Distribution [Vd/F]
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Day 1 (Baseline) and Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
mL
  First dose | 44028.830 (21667.338)
  Last dose | 40693.327 (18934.484)

26. Secondary Outcome: Apparent Clearance [CL/F]
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Day 1 and Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: (mL/hr)
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
(mL/hr)
  First dose (Day 1) | 7064.331 (3062.337)
  Last dose (Week 24) | 6658.927 (3972.114)

27. Secondary Outcome: Minimal or Trough Plasma Concentration [Cmin]
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Week 24 visit at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
ng/mL | 2.321 (1.994)

28. Secondary Outcome: Accumulation Index Calculated as a Ratio of AUCtau (Last Dose)/AUCtau (First Dose)
Description: Pharmacokinetics of Saroglitazar
Time Frame: PK Sampling time points: Day 1 and Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
ratio | 1.134 (0.203)

29. Secondary Outcome: Fluctuation Index
Description: Fluctuation index is the peak trough fluctuation within complete dosing interval at steady state, calculated as PTF (%) = ([Cmax - Cmin]/Cav ) multiplied by 100
Time Frame: PK Sampling time points: Week 24 visits at pre-dose (0), 0.5, 1.0, 2, 3, 4, 6, 8, 10 and 24-hour post-dose
Population: PK population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Saroglitazar Magnesium 4 mg
Number analyzed (Participants) | 6
percentage | 374.965 (182.252)

ADVERSE EVENTS:
Time Frame: 28 Weeks
Arm/Group | Saroglitazar Magnesium 4 mg
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saroglitazar Magnesium 4 mg (N=20)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1
Gastroenteritis viral (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saroglitazar Magnesium 4 mg (N=20)
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Lipase increased (Investigations) | 2
Glomerular filtration rate decreased (Investigations) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Anal incontinence (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Mesenteric artery stenosis (Gastrointestinal disorders) | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Skin neoplasm excision (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03639623/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT03639623/SAP_001.pdf